CLINICAL TRIAL: NCT01204073
Title: A Multicenter, Open-Label, Dose-Escalation, Phase 1 Study of TAK-441, an Oral Hedgehog Signaling Pathway Inhibitor, in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: A Study of TAK-441 in Adult Patients With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C24002; 2010-021311-17 (EudraCT Number)
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Nonhematologic Malignancies; Carcinoma, Basal Cell
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — TAK-441

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-441 (Experimental)
  Interventions: Drug: TAK-441

INTERVENTIONS:
Drug: TAK-441 — TAK-441 will be administered as an oral tablet as follows:
  Patients enrolled in the dose escalation cohorts will receive:
  * A single-dose administration on Day 1, followed by a 1-week washout period during which pharmacokinetics is assessed
  * Continuous daily dosing on Days 8 through 28 in Cycle 1
  * In subsequent cycles, continuous daily dosing over 21 days, repeated continuously
  Patients enrolled in the expansion cohorts will receive continuous daily dosing on Days 1 through 21 of each 21-day cycle

SUMMARY:
This is the first study in which TAK-441 is administered to humans. The patient population will consist of adults aged 18 or older who have advanced nonhematologic malignancies and for whom standard treatment is no longer effective or does not offer curative or life-prolonging potential. Following completion of the dose escalation study, patients will be enrolled as part of 2 expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

* Male or female 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Diagnosis of a nonhematologic malignancy for which standard treatment is no longer effective or does not offer curative or life-prolonging potential
* Meet other clinical, radiographic or laboratory inclusion criteria as specified in the protocol
* Voluntary written consent

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Life-threatening illness unrelated to cancer
* Receiving other treatment (radiotherapy, antineoplastics or investigational agents) within protocol specified windows of first dose of TAK-441
* Patients with brain metastases who do not meet criteria specified in study protocol
* Known history of human immunodeficiency virus (HIV) infection, hepatitis B or hepatitis C
* Major surgery within 14 days before the first dose of TAK-441
* Infection requiring systemic therapy, or other serious infection within 14 days of the first dose of TAK-441
* Do not meet other clinical, laboratory or radiographic criteria as specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-10; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety profile, maximum tolerated dose (MTD) or maximum feasible dose (MFD) of TAK-441 administered as an oral formulation in patients wtih advanced nonhematologic malignancies | From first dose of TAK-441 through 30 days after the last dose of TAK-441
  Adverse events, serious adverse events, dose-limiting toxicities, assessments of clinical laboratory values, electrocardiogram parameters and vital sign measurements

SECONDARY OUTCOMES:
Single-dose and multiple-dose plasma pharmacokinetics (PK) of TAK-441 | Sampling during Cycle 1 (Days 1-28)
  Including but not limited to maximum plasma concentration (Cmax), first time to plasma concentration (Tmax) and area under the plasma concentration versus time curve (AUC)
Pharmacodynamic effect of TAK-441 on Gli 1 expression in skin | Cycle 1 Day 22
Pharmacodynamic effect of TAK-441 on Gli 1 expression in tumors (expansion cohorts only) | Cycle 1 Day 15
Antitumor activity of TAK-441 administered as a single-agent therapy based on investigators' assessments of tumor response in patients who have advanced basal cell carcinoma | Days 15-21 of cycles 2, 4 and every fourth cycle thereafter; and end of study
  Based on the investigator's assessment using the Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (2):
- United States (2):
  - Mayo Clinic, Scottsdale, Arizona
  - Premiere Oncology, A Medical Corporation, Santa Monica, California